CLINICAL TRIAL: NCT06038084
Title: A Prospective, Multi-center, Active-control, Parallel Group, Randomized, Double-blinded, Non-inferiority Investigator Initiative Clinical Trial to Evaluate the Efficacy and Safety of Acute Bronchitis Symptoms Improvement for Bronpass Tab. Compared to Erdos Capsule on Patients With Acute Bronchitis
Brief Title: Evaluate the Efficacy and Safety of Acute Bronchitis Symptoms Improvement for Bronpass Tab. Compared to Erdos Capsule
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kwang-Ha Yoo (Other)
Collaborators: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Kwang-Ha Yoo, Professor, Konkuk University Medical Center
Organization: Konkuk University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL-BRPS-501
Record Dates: First submitted 2023-07-24; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Acute Bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronpass Tab. (Experimental)
  Interventions: Drug: Bronpass Tab.; Drug: Placebo of Erdos capsule
- Erdos capsule (Active Comparator)
  Interventions: Drug: Erdos capsule; Drug: Placebo of Bronpass Tab.

INTERVENTIONS:
Drug: Bronpass Tab. — Twice a day
  Arms: Bronpass Tab.
Drug: Placebo of Erdos capsule — Three times a day (It is for the masking.)
  Arms: Bronpass Tab.
Drug: Erdos capsule — Three times a day
  Arms: Erdos capsule
Drug: Placebo of Bronpass Tab. — Twice a day (It is for the masking.)
  Arms: Erdos capsule

SUMMARY:
The purpose of this clinical trial is to evaluate the acute bronchitis symptom relief effect of Bronpass tab. compared to Erdos capsule, and compare and evaluate the safety.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to evaluate the following in patients with acute bronchitis at the 7th day of administration of the investigational drug.

primary purpose: Prove the non-inferiority of the acute bronchitis symptom relief effect of Bronpass tab. compared to Erdos capsule, and compare and evaluate the safety.

secondary purpose: Compare and evaluate the effect of improving clinical symptoms, including sputum symptoms, of Bronpass tab. compared to Erdos capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 19 to 80 at the time of screening
2. Patients with an acute bronchitis severity score (BSS) of 5 or higher at the time of screening and the first day of administration of the investigational drug
3. Patients with symptoms of acute bronchitis within 48 hours from the time of screening
4. Patients who voluntarily gave written consent to participate in this clinical trial

Exclusion Criteria:

1. Patients with a known hypersensitivity reaction to the components of this investigational product
2. Patients with respiratory and systemic infections requiring systemic antibiotic treatment
3. Patients with clotting disorders or bleeding tendencies
4. Patients with peptic ulcer at the time of screening
5. Severe lung diseases that may affect the efficacy evaluation of this clinical trial at the discretion of the investigator
6. For screening test results, creatinine clearance < 25 mL/min or AST, ALT more than 3 times the upper limit of normal
7. A person who have administered systemic corticosteroids or immunosuppressants within 4 weeks of the first administration of the investigational drug
8. A person who have administered antiviral drugs, systemic/inhaled glucocorticosteroids within 48 hours of the first administration of investigational drugs
9. A person who have administered mucolytics, sputum discharge agents, antitussives, herbal medicines with antitussive/ expectorant effects, and antihistamines within 48 hours of the first administration of investigational drugs
10. A person who need or plan to take contraindicated drugs or therapies during this clinical trial period
11. Patient with liver cirrhosis or cystathionine synthetase deficiency
12. Patient who have clinically significant diseases and disorders in the cardiovascular system, endocrine system, and central nervous system at the time of screening, or who have a history of malignant tumors or mental disorders (eg. depression) (However, participation is possible if there is no recurrence for more than 5 years after surgery at the time of screening)
13. A person with a history of alcoholism or drug abuse
14. Heavy smokers (more than 15 cigarettes per day) within 4 weeks from the time of screening
15. Pregnant or lactating
16. Among female subjects of childbearing potential, women who do not intend to use appropriate contraceptive methods or plan to become pregnant during this clinical trial
17. A person who administered other investigational drugs within 4 weeks from the time of screening
18. A person who are not suitable for participation in this clinical trial under the judgment of the investigator

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Change in BSS(Bronchitis severity score) total score | Visit 3 (Day 7)
  Change in BSS(Bronchitis severity score) total score at 7 days after administration of investigational drug compared to baseline
  * The total BSS score ranges from 0 to 20, with higher scores indicating greater severity of symptoms.

SECONDARY OUTCOMES:
Change in BSS(Bronchitis severity score) score by symptom (cough, sputum, dyspnea, chest pain when coughing, crackles/rhonchus) | Visit 3 (Day 7)
  Change in BSS(Bronchitis severity score) score by symptom (cough, sputum, dyspnea, chest pain when coughing, crackles/rhonchus) at 7 days after administration of the investigational drug compared to baseline
  * The BSS score range for each symptom is 0 to 4 with a higher score indicating a greater severity of symptom.
Overall improvement as assessed by the investigator using the investigator's overall improvement evaluation sheet (5-point scale) | Visit 3 (Day 7)
  Overall improvement judged by the investigator on the treatment response at 7 days after administration of the investigational product
  * The investigator's overall improvement evaluation sheet is a 5-point scale(ranges from 1 to 5) evaluation sheet where a higher score indicates a greater improvement of the subject's symptom.
Satisfaction evaluated by the subject using the subject's satisfaction evaluation sheet (5-point scale) | Visit 3 (Day 7)
  Satisfaction of subjects on the treatment response at 7 days after administration of investigational drug
  * The subject's satisfaction evaluation sheet is a 5-point scale(ranges from 1 to 5) evaluation sheet where a higher score indicates a greater satisfaction.
Number of rescue drug doses | Visit 3 (Day 7)
  Number of rescue drug doses at 7 days after administration of investigational drug
Changes in inflammatory marker (CRP in mg/L) at 7 days after administration of investigational drugs compared to baseline | Visit 3 (Day 7)
  Present the descriptive statistics (Mean, standard deviation, median value, minimum value, maximum value) for the change in inflammatory marker (CRP in mg/L) at 7 days after administration of the investigational drug. And compare the difference in the amount of change between the groups on the 7th day compared to the baseline.
Changes in inflammatory marker (TNF-α in pg/mL) at 7 days after administration of investigational drugs compared to baseline | Visit 3 (Day 7)
  Present the descriptive statistics (Mean, standard deviation, median value, minimum value, maximum value) for the change in inflammatory marker (TNF-α in pg/mL) at 7 days after administration of the investigational drug. And compare the difference in the amount of change between the groups on the 7th day compared to the baseline.
Changes in inflammatory marker (IL-1β in pg/mL) at 7 days after administration of investigational drugs compared to baseline | Visit 3 (Day 7)
  Present the descriptive statistics (Mean, standard deviation, median value, minimum value, maximum value) for the change in inflammatory marker (IL-1β in pg/mL) at 7 days after administration of the investigational drug. And compare the difference in the amount of change between the groups on the 7th day compared to the baseline.
Changes in inflammatory marker (IL-6 in pg/mL) at 7 days after administration of investigational drugs compared to baseline | Visit 3 (Day 7)
  Present the descriptive statistics (Mean, standard deviation, median value, minimum value, maximum value) for the change in inflammatory marker (IL-6 in pg/mL) at 7 days after administration of the investigational drug. And compare the difference in the amount of change between the groups on the 7th day compared to the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Hospital, Seoul, South Korea